CLINICAL TRIAL: NCT00134979
Title: Efficacy and Safety of Formoterol Certihaler, Tiotropium HandiHaler and Tiotropium HandiHaler in Combination With Formoterol Certihaler in Patients With Stable Chronic Obstructive Pulmonary Disease
Brief Title: Formoterol Certihaler, Tiotropium HandiHaler and Tiotropium HandiHaler in Combination With Formoterol Certihaler in Patients With Stable Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CFOR258F2402
Record Dates: First submitted 2005-07-26; First posted 2005-08-25 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD, formoterol,
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Formoterol Fumarate

INTERVENTIONS:
Drug: Formoterol

SUMMARY:
This study is not being conducted in the United States.

This study is designed to provide efficacy and safety data for formoterol 10µg twice-a-day (b.i.d.) delivered by the Certihaler in patients with chronic obstructive pulmonary disease (COPD). This study is also designed to compare the efficacy and safety of therapy with formoterol (Certihaler)10µg b.i.d. added to tiotropium (HandiHaler) 18µg once daily (o.d.) compared with tiotropium (HandiHaler) 18µg o.d. monotherapy, and to compare the safety and efficacy of formoterol 10µg b.i.d. (Certihaler) with tiotropium 18µg o.d. (HandiHaler).

ELIGIBILITY:
Inclusion Criteria:

* Co-operative males or females with a diagnosis of moderate COPD as per the Global Initiative for Chronic Obstructive Lung Disease (GOLD) criteria with an age at onset ≥ 40 years.
* Current or previous smokers with a smoking history of ≥ 10 pack-years. Ten pack-years is defined as 20 cigarettes a day for 10 years, or 10 cigarettes a day for 20 years etc.
* Pre-bronchodilator forced expiratory volume in one second (FEV1) < 70% of patient's predicted normal value and ≥ 1.00 L, with FEV1/forced vital capacity (FVC) < 70% at Visit 2.
* A total symptom score from the patient diary of more than 0 on at least 4 of the last 7 days prior to Visit 3

Exclusion Criteria:

* Pregnant women, nursing mothers, and females of childbearing potential, regardless of whether or not sexually active, who do not use a reliable contraceptive method (oral, mechanical, subcutaneous or surgical contraception).
* Patients who have been hospitalized for an acute exacerbation of their airway diseases in the month prior to Visit 1 or during screening.
* Patients who have had a respiratory tract infection within 1 month prior to Visit 1. Patients who develop a respiratory tract infection during the screening period must discontinue from the trial, but will be permitted to re-enroll at a later date (at least 1 month after the resolution of the respiratory tract infection).
* Patients with concomitant pulmonary disease including a history of cancer (all), pulmonary tuberculosis or congenital bronchiectasis.
* History of asthma

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 847 (Actual)
Dates: Start 2004-10; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Forced Expiratory Volume in 1 second measured at 2 h post dosing following 24 weeks treatment

SECONDARY OUTCOMES:
Forced Expiratory Volume in 1 second measured pre-dose, 5 minutes, 2 h and 3 h post dose at day 1, week 12 and week 24
Forced Vital Capacity measured pre-dose, 5 minutes, 2 h and 3 h post dose at day 1, week 12 and week 24
St. George's Respiratory Questionnaire following 12 and 24 weeks of treatment.
COPD "Bad Days" recorded throughout study
COPD "Exacerbation days" recorded throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (1):
- Novartis Pharma AG, Switzerland

REFERENCES:
- [Derived] Vogelmeier C, Kardos P, Harari S, Gans SJ, Stenglein S, Thirlwell J. Formoterol mono- and combination therapy with tiotropium in patients with COPD: a 6-month study. Respir Med. 2008 Nov;102(11):1511-20. doi: 10.1016/j.rmed.2008.07.020. Epub 2008 Sep 19. PMID 18804362